CLINICAL TRIAL: NCT04584905
Title: Nutritional Assessment of Children With Chronic Kidney Disease Attending Assuit University Children Hospital
Brief Title: Nutritional Assessment of Children With Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maram Mohamed Amir Fathy, principal investigator, Assiut University
Other Study IDs: nutrition in CKD
Record Dates: First submitted 2020-09-23; First posted 2020-10-14 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Nutrition Disorders, Child
Keywords: chronic kidney disease
MeSH Terms: conditions — Child Nutrition Disorders; Renal Insufficiency, Chronic | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: dietary supplements for CKD patients — follow up and assessment of nutritional status of CKD patients

SUMMARY:
Primary outcome is assessment of nutritional status of children with CKD. Secondary outcome is assessment STAMP screening tool for detection of malnutrition of CKD children.

DETAILED DESCRIPTION:
Pediatric Chronic Kidney Disease (CKD) has systemic implication on all aspects of normal development, including nutrition, growth, bone and mineral metabolism and neurocognitive function .

Chronic Kidney Disease (CKD) introduces a unique set of nutritional challenges for the growing and developing child .

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes.
* Diagnosed as chronic kidney disease.
* Age: 2 years up to 15 Years Children.

Exclusion Criteria:

* • Age: less than 2 years old child and more than 15 years old child.

  * Previously diagnosed to have any co- morbid or systemic disease other than CKD.
  * Irregular dialysis.
  * Renal transplant.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children of both sexes. Diagnosed as chronic kidney disease. Age: 2 years up to 15 Years Children
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of nutritional status of children with CKD. | from January 2021 to June 2021
  by measuring body mass index in kg/m2.

SECONDARY OUTCOMES:
Assess STAMP screening tool | from January 2021 to June 2021
  Five steps STAMP assessment for detection of malnutrition in children with CKD.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Universty Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No